CLINICAL TRIAL: NCT00096265
Title: A Phase III Trial Comparing Whole Brain Radiation and Stereotactic Radiosurgery Alone Versus With Temozolomide or Erlotinib in Patients With Non-Small Cell Lung Cancer and 1-3 Brain Metastases
Brief Title: Radiation Therapy and Stereotactic Radiosurgery With or Without Temozolomide or Erlotinib in Treating Patients With Brain Metastases Secondary to Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00720; NCI-2009-00720 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000389490; RTOG 0320; RTOG 0320 (Other: Radiation Therapy Oncology Group); RTOG-0320 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Erlotinib Hydrochloride; Radiosurgery; Temozolomide

ARMS (3):
- Arm I (Active Comparator): Patients undergo whole brain radiotherapy (WBRT) once daily on days 1-5, 8-12, and 15-19. Within 14 days after completion of WBRT, patients undergo stereotactic radiosurgery.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Stereotactic Radiosurgery
- Arm II (Experimental): Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral temozolomide once daily on days 1-21. Beginning 4 weeks after completion of WBRT, patients may receive oral temozolomide alone once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Stereotactic Radiosurgery; Drug: Temozolomide
- Arm III (Experimental): Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral erlotinib once daily for up to 6 months.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Erlotinib Hydrochloride; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Patients undergo radiation therapy once daily for approximately 3 weeks
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Drug: Erlotinib Hydrochloride — Given orally
  Other Names: Cp-358,774; OSI-774; Tarceva
  Arms: Arm III
Radiation: Stereotactic Radiosurgery — Patients undergo surgery after radiation therapy
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Drug: Temozolomide — Given orally
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac
  Arms: Arm II

SUMMARY:
This randomized phase III trial is studying whole-brain radiation therapy and stereotactic radiosurgery with or without temozolomide or erlotinib to see how well they work compared to whole-brain radiation therapy and stereotactic radiosurgery in treating patients with brain metastases secondary to non-small cell lung cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Stereotactic radiosurgery may be able to deliver x-rays directly to the tumor and cause less damage to normal tissue. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by blocking blood flow to the tumor. It is not yet known whether radiation therapy and stereotactic radiosurgery are more effective with or without temozolomide or erlotinib in treating brain metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare survival in patients with non-small cell lung cancer and brain metastases treated with whole brain radiotherapy and stereotactic radiosurgery with vs without temozolomide or erlotinib.

SECONDARY OBJECTIVES:

I. Compare time to CNS progression in patients treated with these regimens. II. Compare quality-adjusted survival in patients treated with these regimens. III. Compare 3-month quality of life in patients treated with these regimens. IV. Compare the 6-month performance status of patients treated with these regimens.

V. Compare 6-month steroid dependence in patients treated with these regimens. VI. Compare cause of death (neurologic vs other) in patients treated with these regimens.

VII. Determine the effects of non-protocol chemotherapy in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age and the presence of extracranial metastases (< 65 years old AND no extracranial metastases vs ≥ 65 years old OR extracranial metastases), number of metastases (1 vs 2 or 3), and extent of extracranial disease (none vs present). Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients undergo whole brain radiotherapy (WBRT) once daily on days 1-5, 8-12, and 15-19. Within 14 days after completion of WBRT, patients undergo stereotactic radiosurgery.

ARM II: Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral temozolomide once daily on days 1-21. Beginning 4 weeks after completion of WBRT, patients may receive oral temozolomide alone once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM III: Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral erlotinib once daily for up to 6 months.

In all arms, patients with recurrent brain metastases may undergo additional stereotactic radiosurgery.

Quality of life is assessed at baseline and at 3, 6, 9, 12, 18, and 24 months.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* One to 3 intraparenchymal brain metastases by contrast-enhanced MRI, meeting the following criteria:

  * Well circumscribed tumor(s)
  * Maximum diameter ≤ 4.0 cm

    * If multiple lesions are present and one lesion is at the maximum diameter, the other lesions must not exceed 3.0 cm in maximum diameter
  * No metastases within 10 mm of the optic apparatus such that a portion of the optic nerve or chiasm would be included in the high-dose stereotactic radiosurgery boost field
  * No metastases in the brainstem, midbrain, pons, or medulla
* No prior complete resection of all known brain metastases

  * Subtotal resection allowed provided residual disease is ≤ 4.0 cm in maximum diameter
* No clinical or radiographic evidence of progression (other than study lesion[s]) within the past month

  * Patients with brain metastases at initial presentation do not require 1 month of scans documenting stable disease
* Stable extracranial metastases allowed

  * No known or pre-existing liver metastases
* No leptomeningeal metastases by MRI or cerebrospinal fluid evaluation
* Synchronous brain metastases at initial diagnosis allowed
* Performance status - Zubrod 0-1
* Hemoglobin ≥ 8 g/dL
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* AST < 2 times upper limit of normal (ULN)
* Alkaline phosphatase < 2 times ULN unless due to elevated bone metastases
* Total bilirubin normal
* Lactic dehydrogenase < 2 times ULN
* Creatinine < 1.5 times ULN
* No clinically active interstitial lung disease

  * Chronic stable asymptomatic radiographic changes allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Neurologic function status 0-2
* No other major medical illness or psychiatric impairment that would preclude study participation
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to erlotinib or temozolomide
* No concurrent immunotherapy
* No concurrent biologic therapy, excluding growth factors and epoetin alfa
* No prior temozolomide or erlotinib
* No other concurrent chemotherapy during study radiotherapy

  * Other concurrent chemotherapy allowed after study radiotherapy, except for the following:

    * Temozolomide or erlotinib (arm I only)
    * Erlotinib (arm II only)
    * Temozolomide (arm III only)
* No prior cranial radiotherapy
* No concurrent intensity-modulated radiotherapy
* Concurrent radiotherapy to painful bone lesions allowed

  * No concurrent radiotherapy to more than 15% of bone marrow
* No other concurrent therapy for brain metastases unless a recurrence is detected
* More than 30 days since prior investigational drugs
* No concurrent enzyme-inducing antiepileptic drugs including, but not limited to, any of the following (for patients randomized to receive erlotinib):

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Phenobarbital
  * Primidone
  * Oxcarbazepine
* No other concurrent investigational drugs
* No concurrent Hypericum perforatum (St. John's wort)
* No drugs that alter gastric pH (e.g., proton pump inhibitors or H2 antagonists) within 4 hours after erlotinib administration (arm III patients only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-10-06 (Actual); Primary Completion 2011-06-14 (Actual); Study Completion 2012-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sperduto, Principal Investigator — Radiation Therapy Oncology Group
Locations (83):
- United States (80):
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Scottsdale Health Care-Osborn, Scottsdale, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Bay Medical Center, Panama City, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Saint Margaret Health-Hammond Campus, Hammond, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Finley Hospital, Dubuque, Iowa
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - University of Rochester, Rochester, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Radiation Therapy Oncology Group, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
- Canada (3):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Ottawa Hospital-Civic Campus, Ottawa, Ontario
  - McGill University Department of Oncology, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- WBRT + SRS: Patients undergo whole brain radiotherapy (WBRT) once daily on days 1-5, 8-12, and 15-19. Within 14 days after completion of WBRT, patients undergo stereotactic radiosurgery.
- Temozolomide + WBRT + SRS: Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral temozolomide once daily on days 1-21. Beginning 4 weeks after completion of WBRT, patients may receive oral temozolomide alone once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Erlotinib + WBRT + SRS: Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral erlotinib once daily for up to 6 months.
Period: Overall Study
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Started | 45 | 40 | 41
Completed | 44 (Subjects contributing data to the primary analysis are considered to have completed the study.) | 40 | 41
Not Completed | 1 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS | Total
Number analyzed (Participants) | 45 | 40 | 41 | 126
Age, Continuous [Median (Full Range); unit: years] | 63 [42 to 89] | 63 [39 to 83] | 61 [46 to 85] | 63 [39 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 18 | 58
  Male | 23 | 22 | 23 | 68

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival time is defined as time from randomization to date of death from any cause and estimated by the Kaplan-Meier method. Patients last known to be alive are censored at date of last contact.
Time Frame: From randomization to date of death or last follow-up, up to 48.1 months. Analysis occurs after all patients have been potentially followed for 9 months.
Population: All eligible patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Number analyzed (Participants) | 44 | 40 | 41
months | 13.4 [6.5 to 20.8] | 6.3 [3.4 to 10.1] | 6.1 [3.6 to 12.1]
Statistical Analysis 1: Comparison: WBRT + SRS vs Temozolomide + WBRT + SRS; 120 patients per arm required to detect a 33% reduction in hazard rate corresponding to improvement in MST of 5.9 (null hypothesis) to 8.9 months with a one-sided type I error rate of 0.025 and 85% power; Test type: Superiority or Other; p = 0.93, Log Rank — One-sided; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.89 to 2.31] — WBRT + SRS is the denominator of the hazard ratio
Statistical Analysis 2: Comparison: WBRT + SRS vs Erlotinib + WBRT + SRS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.95, Log Rank — One-sided; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.92 to 2.36] — WBRT + SRS is the denominator of the hazard ratio

2. Secondary Outcome: Rate of CNS Progression (One Year)
Description: CNS progression is defined as any increase in perpendicular bi-dimensional tumor area for any of the 1-3 tracked brain metastases, by any amount, or the appearance of any new brain metastasis on a follow-up MRI (SRS planning scan will not be used to evaluate CNS progression). For lesions smaller than 1 cm in maximum diameter, a maximum increase of 50% in perpendicular bi-dimensional treatment area is necessary to score as progression. This caveat is included to account for potential variability in measurement, which is most susceptible to proportionate errors at smaller sizes. For greater than 1 cm lesions, the definition uses a 25% rule for change. Rates of CNS progression estimated by the cumulative incidence method, with death treated as a competing risk.
Time Frame: From randomization to last follow-up, up to 48.1 months. Analysis occurs after all patients have been potentially followed for 9 months.
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Number analyzed (Participants) | 44 | 40 | 41
percentage of participants | 34.1 [19.8 to 48.4] | 47.4 [31.0 to 63.8] | 27.4 [13.2 to 41.5]
Statistical Analysis 1: Comparison: WBRT + SRS vs Temozolomide + WBRT + SRS; Test type: Superiority; p = 0.30, Gray's test
Statistical Analysis 2: Comparison: Temozolomide + WBRT + SRS vs Erlotinib + WBRT + SRS; Test type: Superiority; p = 0.48, Gray's test

3. Secondary Outcome: Quality-adjusted Survival as Measured by EuroQol 5-dimension Instrument
Description: Quality-adjusted life years (QALY) incorporate the societal-based utilities of health states into expected life years for a health condition. The QALY model is QALY(h,y) where h is a health state and y is the years of life. Higher quality-adjusted life year values represent a better outcome. A patient's health state will be determined from the index score of the EQ-5D-5L patient questionnaire.The EQ-5D-5L is a 2-part self-assessment questionnaire, a 5-item index score and a visual analogue scale, but only the index score is used for quality-adjusted survival. The index score has 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 5 problem levels (1-none to 5-extreme). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state).
Time Frame: as for outcome 2
Population: Eligible patients with any follow-up EQ-5D
Measure: Mean (Standard Deviation); unit: Quality-adjusted life years
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Number analyzed (Participants) | 24 | 19 | 18
Quality-adjusted life years | 16.9 (9.6) | 15.9 (12.0) | 14.4 (12.5)

4. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-Brain (FACT-Br) Score at 3 Months
Description: The Functional Assessment of Cancer Therapy-Brain (FACT-Br) is a 19-item self-report instrument designed to measure multidimensional quality of life in patients with brain cancer. It is to be administered with the FACT-General. There are 5 responses options, with 0=Not a lot and 4=Very much. All items are added together to obtain a total score, which ranges from 0 to 76. Certain items must be reversed before it is added by subtracting the response from 4. It requires at least 50% of the items to be completed while the overall response rate of the FACT-Br including the FACT-G must be greater than 80%. If items are missing, the subscale scores can be prorated. A higher score indicates better QOL. A change of 5 points will be considered a minimal clinically meaningful change. Change from baseline at three months (3 month score - baseline score) will be categorized as improvement if increased, stable if no change, or deterioration if decreased.
Time Frame: From randomization to three months.
Population: Eligible patients with both baseline and 3 month data
Measure: Count of Participants; unit: Participants
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Number analyzed (Participants) | 26 | 16 | 17
Participants
  Deterioration/Decrease | 12 | 10 | 11
  Stable | 8 | 2 | 6
  Improvement/Increase | 6 | 4 | 1
Statistical Analysis 1: Comparison: WBRT + SRS vs Temozolomide + WBRT + SRS; With 70 patients per arm, a 0.05 level chi-square test would have 80% power to distinguish between two groups when the proportions in the three categories are as follows for standard vs. experimental arm, respectively: 25% vs. 50% improvement, 55% vs. 40% stable, and 20% vs. 10% deterioration, or any distribution that corresponds to an effect size, Δ² = Σ(π2j-π1j)2/[2(π2j-π1j)], of 0.0702; Test type: Superiority; p = 0.39, Chi-squared
Statistical Analysis 2: Comparison: WBRT + SRS vs Erlotinib + WBRT + SRS; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.28, Chi-squared

5. Secondary Outcome: Change in Performance Status at Six Months
Description: Compared between two treatment arms using a two-group chi-squared test. Zubrod score will be collected at baseline and follow-up. The Zubrod performance score runs from 0 to 5, with 0 denoting perfect health and 5 death. Change from baseline is calculated as 6-month value - baseline value. Patients with a baseline score who have died by six months will be included in the analysis with a score of 5 at six months.
Time Frame: From randomization to six months.
Population: Eligible patients with baseline and 6 month data
Measure: Count of Participants; unit: Participants
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Number analyzed (Participants) | 40 | 35 | 35
Participants
  Improvement (decrease) | 0 | 1 | 3
  Stable (no change) | 19 | 4 | 2
  Deterioration (increase) | 21 | 30 | 30
Statistical Analysis 1: Comparison: WBRT + SRS vs Temozolomide + WBRT + SRS; 108 with three month performance status data, per arm, would result in a 0.050 level chi-square test with 90% power to distinguish between the groups when the proportions in the 3 categories are characterized by an effect size, Δ² = Σ(π2j-π1j)2/[2(π2j-π1j)], of 0.0586; Test type: Superiority; p = 0.002, Chi-squared
Statistical Analysis 2: Comparison: WBRT + SRS vs Erlotinib + WBRT + SRS; 108 cases with three month performance status data, per arm, would result in a 0.050 level chi-square test with 90% power to distinguish between the groups when the proportions in the 3 categories are characterized by an effect size, Δ² = Σ(π2j-π1j)2/[2(π2j-π1j)], of 0.0586; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: Change in Steroid Dependence at Six Months
Description: Daily steroid dose will be collected at baseline and follow-up, as one of the following: 0-4 mg, >4 to ≤ 8 mg, >8 to ≤12 mg, and >12 mg. Change from baseline at six months will be evaluated to have decreased, remained stable, or increased, based on these categories.
Time Frame: From randomization to six months.
Population: Eligible patients with both baseline and 6 month steroid dose
Measure: Count of Participants; unit: Participants
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Number analyzed (Participants) | 26 | 18 | 17
Participants
  Decrease | 12 | 10 | 10
  Stable | 10 | 4 | 6
  Increase | 4 | 4 | 1
Statistical Analysis 1: Comparison: WBRT + SRS vs Temozolomide + WBRT + SRS; Test type: Superiority — Assuming the survival rate of the standard arm (MST = 5.9 months), then 49% of patients were expected to be alive at six months. Assuming steroid data would be available for 90% of these patients, results in a projection of 52 cases/arm with steroid data at 6 months. With this sample size, a two-sided 0.050 alpha test will have 90% power to distinguish between the groups when the proportions in the 3 categories are characterized by an effect size, Δ² = Σ(π2j-π1j)2/[2(π2j-π1j)], of 0.1217; p = 0.51, Chi-squared
Statistical Analysis 2: Comparison: WBRT + SRS vs Erlotinib + WBRT + SRS; Assuming the survival rate of the standard arm (MST = 5.9 months), then 49% of patients were expected to be alive at six months. Assuming steroid data would be available for 90% of these patients, results in a projection of 52 cases/arm with steroid data at 6 months. With this sample size, a two-sided 0.050 alpha test will have 90% power to distinguish between the groups when the proportions in the 3 categories are characterized by an effect size, Δ² = Σ(π2j-π1j)2/[2(π2j-π1j)], of 0.1217; Test type: Superiority; p = 0.56, Chi-squared

7. Secondary Outcome: Cause of Death (Neurologic vs Other)
Description: Patients were considered to have died neurologic deaths (coded as "Brain Metastases") if they had stable systemic disease and progressive neurologic disease consisting of expanding intracranial masses, CNS hemorrhages, hydrocephalus resulting in herniation or fulminant meningeal carcinomatosis.
Time Frame: as for outcome 2
Population: Eligible patients who died
Measure: Count of Participants; unit: Participants
Arm/Group | WBRT + SRS | Temozolomide + WBRT + SRS | Erlotinib + WBRT + SRS
Number analyzed (Participants) | 35 | 34 | 36
Participants
  Neuroligic death | 6 | 5 | 7
  Other | 29 | 29 | 29
Statistical Analysis 1: Comparison: WBRT + SRS vs Temozolomide + WBRT + SRS; A two group chi-square test with a 0.05 two-sided significance level would have 89% power to detect the difference between a proportion of 0.50 and a proportion of 0.30, or equivalently, of 0.70, when the sample size in each group is 120; Test type: Superiority; p = 0.78, Chi-squared
Statistical Analysis 2: Comparison: WBRT + SRS vs Erlotinib + WBRT + SRS; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.80, Chi-squared

ADVERSE EVENTS:
Description: Per the protocol, toxicity data was collected via CTC 3.0 then mapped to CTCAE 4.0 for reporting on this website. Subjects experiencing more than one of a given adverse event (AE) are counted only once for that AE.
Groups:
- WBRT+SRS: Patients undergo whole brain radiotherapy (WBRT) once daily on days 1-5, 8-12, and 15-19. Within 14 days after completion of WBRT, patients undergo stereotactic radiosurgery. [Data is reported for eligible patients with adverse event information, which is 44 patients.]
- Temozolomide+WBRT+SRS: Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral temozolomide once daily on days 1-21. Beginning 4 weeks after completion of WBRT, patients may receive oral temozolomide alone once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. [Data is reported for eligible patients with adverse event information, which is 39 patients.]
- Erlotinib+WBRT+SRS: Patients undergo WBRT and stereotactic radiosurgery as in arm I. Beginning on the first day of WBRT, patients receive oral erlotinib once daily for up to 6 months. [Data is reported for eligible patients with adverse event information, which is 41 patients.]
Arm/Group | WBRT+SRS | Temozolomide+WBRT+SRS | Erlotinib+WBRT+SRS
Serious Adverse Events (participants affected / at risk) | 10/44 | 22/39 | 12/41
Other Adverse Events (participants affected / at risk) | 28/44 | 32/39 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT+SRS (N=44) | Temozolomide+WBRT+SRS (N=39) | Erlotinib+WBRT+SRS (N=41)
Anemia (Blood and lymphatic system disorders) | 2 | 5 | 4
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Death NOS (General disorders) | 3 | 2 | 2
Edema limbs (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2
Fever (General disorders) | 0 | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Sudden death NOS (General disorders) | 1 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 2 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 1
GGT increased (Investigations) | 0 | 0 | 1
INR increased (Investigations) | 0 | 1 | 0
Investigations - Other (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 4 | 2
Weight loss (Investigations) | 0 | 1 | 2
White blood cell decreased (Investigations) | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 3 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT+SRS (N=44) | Temozolomide+WBRT+SRS (N=39) | Erlotinib+WBRT+SRS (N=41)
Anemia (Blood and lymphatic system disorders) | 7 | 12 | 11
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 3 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 2 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 2 | 2
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 2 | 1 | 0
Blurred vision (Eye disorders) | 1 | 3 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 3
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 1
Eye disorders - Other (Eye disorders) | 1 | 1 | 3
Eye pain (Eye disorders) | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 0 | 0
Watering eyes (Eye disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 10 | 10
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 14
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 2 | 3
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 4 | 2
Nausea (Gastrointestinal disorders) | 7 | 13 | 15
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 7 | 8
Chills (General disorders) | 1 | 0 | 1
Edema face (General disorders) | 2 | 0 | 1
Edema limbs (General disorders) | 2 | 5 | 2
Fatigue (General disorders) | 20 | 24 | 22
Fever (General disorders) | 0 | 1 | 2
Gait disturbance (General disorders) | 1 | 3 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 5
Pain (General disorders) | 0 | 2 | 0
Immune system disorders - Other (Immune system disorders) | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 5 | 5
Lung infection (Infections and infestations) | 2 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Salivary gland infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 10 | 4
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 1 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 4 | 8
Alkaline phosphatase increased (Investigations) | 3 | 4 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 10
Blood bilirubin increased (Investigations) | 0 | 0 | 4
Creatinine increased (Investigations) | 0 | 1 | 3
Fibrinogen decreased (Investigations) | 0 | 2 | 0
GGT increased (Investigations) | 3 | 1 | 3
INR increased (Investigations) | 0 | 4 | 3
Investigations - Other (Investigations) | 0 | 3 | 2
Lymphocyte count decreased (Investigations) | 1 | 2 | 3
Neutrophil count decreased (Investigations) | 1 | 2 | 5
Platelet count decreased (Investigations) | 2 | 7 | 4
Weight gain (Investigations) | 2 | 1 | 0
Weight loss (Investigations) | 3 | 8 | 11
White blood cell decreased (Investigations) | 2 | 3 | 4
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 7 | 13 | 18
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 7 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 5 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 6 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 5 | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Arachnoiditis (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 3 | 4 | 4
Central nervous system necrosis (Nervous system disorders) | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 4 | 4 | 6
Dysgeusia (Nervous system disorders) | 2 | 4 | 8
Dysphasia (Nervous system disorders) | 2 | 2 | 2
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 8 | 7
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 | 0
Ischemia cerebrovascular (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 5 | 2 | 6
Myelitis (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 2 | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 4 | 6 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2 | 5
Pyramidal tract syndrome (Nervous system disorders) | 0 | 2 | 0
Seizure (Nervous system disorders) | 2 | 4 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Tremor (Nervous system disorders) | 1 | 2 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2 | 2
Confusion (Psychiatric disorders) | 4 | 2 | 6
Depression (Psychiatric disorders) | 2 | 1 | 4
Insomnia (Psychiatric disorders) | 3 | 5 | 4
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Personality change (Psychiatric disorders) | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 2
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 3 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 11 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 3
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 3 | 1
Thromboembolic event (Vascular disorders) | 2 | 3 | 1
Vascular disorders - Other (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 126 subjects accrued out of 381 planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less